CLINICAL TRIAL: NCT04888988
Title: Multi-Center Randomized Controlled Phase II Trial of Exercise to Treat Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Testing the Effects of Exercise on Chemotherapy-Induced Peripheral Neuropathy
Acronym: CIPN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Po-Ju Lin, URCC Study Co-Chair, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: URCC19075; R21CA256154 (NIH); UG1CA189961 (NIH); NCI-2020-11456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC19075 (Other: University of Rochester NCORP Research Base); URCC-19075 (Other: DCP); URCC-19075 (Other: CTEP)
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Magnetic Resonance Spectroscopy; Restraint, Physical

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (EXCAP, tactile sensitivity test, counseling) (Experimental): Participants undergo the EXCAP intervention consisting of a home-based, self-directed, individually tailored progressive walking and resistance program for up to 6 weeks. Participants also undergo a tactile sensitivity test at baseline and after completion of EXCAP over 15-25 minutes. In addition, participants meet with a certified exercise instructor over 45 minutes at baseline and 2 additional booster meetings over 15-30 minutes during weeks 2 and 3 or weeks 4 and 5. Participants may optionally undergo MRI on study.
  Interventions: Other: Exercise Counseling; Other: Exercise Intervention; Procedure: Magnetic Resonance Imaging; Other: Neuropathy Assessment; Other: Questionnaire Administration
- Arm 2 (usual care, tactile sensitivity test) (Active Comparator): Participants receive usual care for 6 weeks. At the end of the study, participants may receive the exercise kit and complete the EXCAP program as in Arm 1. Participants also undergo a tactile sensitivity test at baseline and after completion of EXCAP over 15-25 minutes. Participants may optionally undergo MRI on study.
  Interventions: Other: Best Practice; Other: Exercise Counseling; Other: Exercise Intervention; Procedure: Magnetic Resonance Imaging; Other: Neuropathy Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm 2 (usual care, tactile sensitivity test)
Other: Exercise Counseling — Meet with certified exercise instructor
Other: Exercise Intervention — Participate in the EXCAP program
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Neuropathy Assessment — Undergo tactile sensitivity test
  Other Names: Assessment for Neuropathic Pain
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies whether using exercise is better than the usual approach for treating chemotherapy-induced peripheral neuropathy (CIPN). CIPN occurs when chemotherapy damages the nerves communicating between the brain, spinal cord, and the rest of the body. The usual approach for treating CIPN is treatment with drugs that help reduce symptoms of other types of neuropathy (for example, from diabetes). However, these drugs do not treat all symptoms of CIPN. Exercise may help to reduce CIPN symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the preliminary efficacy of exercise versus (vs.) standard care for treating CIPN (via patient-reported CIPN-20 total score).

SECONDARY OBJECTIVES:

I. Assess the preliminary efficacy of exercise vs. standard care on individual symptoms of CIPN (via CIPN Symptom Inventory; i.e., numbness, tingling, burning/shooting pain, and cramping in the hands and feet).

II. Assess the preliminary efficacy of exercise vs. standard care on a clinical test of CIPN symptoms (via the tactile sensitivity in the fingers and toes).

III. Assess the effects of exercise vs. standard care on two possible CIPN mechanisms, namely interoception (via Multidimensional Assessment of Interoceptive Awareness version 2 [MAIA-2] questionnaire).

EXPLORATORY OBJECTIVES:

I. Assess the effects of exercise vs. standard care on other common symptoms related to cancer, chemotherapy, and CIPN, including:

Ia. Daily Diary of symptoms of CIPN. Ib. An array of cancer and treatment symptoms (MD Anderson Symptom Inventory; MDASI).

Ic. Anxiety and depression (hospital anxiety and depression scale; HADS). Id. Pain catastrophizing (pain catastrophizing scale; PCS). Ie. Cognitive impairment (Functional Assessment of Cancer Therapy-Cognitive [FACT-Cog]).

If. Fatigue (brief fatigue inventory; BFI). Ig. Quality of life (Functional Assessment of Cancer Therapy - General [FACT-G]).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM 1 (EXERCISE): Participants undergo the exercise for cancer patients (EXCAP) intervention consisting of a home-based, self-directed, individually tailored progressive walking and resistance program for up to 6 weeks. Participants also undergo a tactile sensitivity test at baseline and after completion of EXCAP over 15-25 minutes. In addition, participants meet with a certified exercise instructor over 45 minutes at baseline and 2 additional booster meetings over 15-30 minutes during weeks 2 and 3 or weeks 4 and 5.

ARM 2 (CONTROL): Participants receive usual care for 6 weeks. At the end of the study, participants may receive the exercise kit and complete the EXCAP program as in Arm 1. Participants also undergo a tactile sensitivity test at baseline and after completion of EXCAP over 15-25 minutes.

Participants may optionally undergo magnetic resonance imaging (MRI) on study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer
* Have received neurotoxic chemotherapy within the past nine months (could still be on chemotherapy or have already completed chemotherapy; i.e., taxane-, platinum-, vinca alkaloid-, epothilone-, or proteasome inhibitor-based chemotherapy
* Report one or more symptoms of CIPN at a level of >= 4 on the CIPN symptom inventory on the Screening Form
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Have at least six months life expectancy
* Be at least 18 years of age
* Be able to read and understand English
* Be able to provide written informed consent

Exclusion Criteria:

* Have physical limitations (e.g., cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in a low to moderate intensity home-based walking and progressive resistance exercise program, according to the participant's physician (e.g., oncologist, primary care) or physician's designee
* Be identified as in the active or maintenance stage of exercise behavior per the Exercise Stages of Change Question on the Screening Form
* Have planned surgery or radiation treatment during the course of the study (hormonal and biologic therapy is allowed)
* Have contraindications for MRI scanning, per the MRI safety screening procedures of the MRI facility to be utilized for this participant
* Are pregnant of have plans to become pregnant during the course of the study. Documentation of pregnancy and use of contraception can be obtained from the medical record.
* Have a current or prior cancer in the central nervous system (spine, brainstem, brain) as this would interfere with assessments of brain functional connectivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-induced peripheral neuropathy (CIPN) symptom severity | Week 6 post randomization
  Will estimate the effects of exercise versus usual care on CIPN using analysis of covariance (ANCOVA). Will be measured by the mean European Organization for Research and Treatment of Cancer-CIPN20. The model will include CIPN-20 at Week 6 as the outcome, treatment group (exercise vs. usual care) as the independent variable of interest and the pre-intervention CIPN-20 score as a covariate.

SECONDARY OUTCOMES:
Effects of exercise on the severity of CIPN symptoms | Up to 6 weeks post randomization
  We will estimate the effects of exercise vs. usual care on CIPN symptoms (i.e., hot/burning or sharp/shooting pain in the hands or feet, numbness or tingling in the hands or feet) collected from the daily symptom inventory (0-10 severity) using analysis of covariance (ANCOVA). The model will include the average of daily symptom inventory for each CIPN symptom at post-intervention as the outcome, controlling for the average of daily symptom inventory for each CIPN symptom at pre-intervention.
Effects of exercise on tactile sensitivity | Up to 6 weeks post randomization
  We will estimate the effects of exercise vs. usual care on tactile sensitivity in the fingers and toes, assessed via an established touch test procedure with a set of monofilaments, using analysis of covariance (ANCOVA). The model will include the tactile sensitivity score at post-intervention as the outcome, controlling for the pre-intervention score.
Effect of exercise on interoception | Up to 6 weeks post randomization
  We will estimate the effects of exercise vs. usual care on interoception, measured via the Multidimensional Assessment of Interoceptive Awareness version 2 (MAIA-2), using analysis of covariance (ANCOVA). The model will include the MAIA-2 total score at post-intervention as the outcome, controlling for the pre-intervention MAIA-2 total score.

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Kleckner, Principal Investigator — University of Rochester NCORP Research Base
Locations (93):
- United States (93):
  - Kaiser Permanente-Fresno, Fresno, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - SIH Cancer Institute, Carterville, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Lake Regional Hospital, Osage Beach, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - CaroMont Health - Lincoln Cancer Center, Lincolnton, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Nash UNC HealthCare, Rocky Mount, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Chesapeake Regional Medical Center, Chesapeake, Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin